CLINICAL TRIAL: NCT02416934
Title: The Effects of Perioperative Steroids on Dysphagia Following Anterior Cervical Spine Surgery: A Randomized, Prospective, Double-Blind Study.
Brief Title: Dysphagia Following Anterior Cervical Spine Surgery; Steroid vs Saline
Acronym: DysDexVSSal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Sanford E Emery, MD, MBA, Professor and Chair West Virginia University Department of Orthopaedics, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1405296745
Record Dates: First submitted 2015-01-09; First posted 2015-04-15 (Estimated); Results first posted 2018-03-30 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Dexamethasone; Steroids; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment 1; Dexamethasone (Experimental): Patients undergoing elective anterior cervical spine surgery will be seen by spine surgeons. After consent the Bazaz and Dysphagia Short Questionnaire will be administered at baseline prior to surgery, Day 1, Day 2, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  Patients will be randomized to either the steroid administration group or the saline administration group. Patients randomized to the experimental (steroid) group will receive 0.3 mg/kg of intravenous dexamethasone within one hour of the incision, then 0.15 mg/kg every eight hours for two doses. This dosage is approximately 20 mg, 10 mg, and 10 mg of dexamethasone. Patients in the control(saline) group will receive a similar volume of saline on the same schedule for three doses.
  Interventions: Drug: Treatment 1; Dexamethasone
- Treatment 0; Saline placebo (Placebo Comparator): Patients undergoing elective anterior cervical spine surgery will be seen by spine surgeons. After consent the Bazaz and Dysphagia Short Questionnaire will be administered at baseline prior to surgery, Day 1, Day 2, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  Patients will be randomized to either the steroid administration group or the saline administration group. Patients randomized to the experimental (steroid) group will receive 0.3 mg/kg of intravenous dexamethasone within one hour of the incision, then 0.15 mg/kg every eight hours for two doses. This dosage is approximately 20 mg, 10 mg, and 10 mg of dexamethasone. Patients in the control(saline) group will receive a similar volume of saline on the same schedule for three doses.
  Interventions: Drug: Treatment 0; Saline placebo

INTERVENTIONS:
Drug: Treatment 1; Dexamethasone — Dexamethasone IV given within the first hour of surgery; second dose given 8 hours after first dose; third dose given 8 hours after second dose.
  Other Names: Steroid
  Arms: Treatment 1; Dexamethasone
Drug: Treatment 0; Saline placebo — Saline (placebo) IV given within the first hour of surgery; second dose given 8 hours after first dose; third dose given 8 hours after second dose.
  Other Names: Saline
  Arms: Treatment 0; Saline placebo

SUMMARY:
This prospective, randomized, double blind, controlled study evaluates the effect of perioperative IV steroids versus saline on swallowing after anterior cervical spine surgery.

DETAILED DESCRIPTION:
This investigation is a prospective, randomized, double-blind, controlled trial testing peri-operative steroids versus saline and the effect on swallowing after anterior cervical spine surgery. Swallowing symptoms will be measured using the patient reported Bazaz (Bazaz) scale and the Dysphagia Short Questionnaire (DSQ). Swallowing data will be obtained pre-operatively, one day and two days post-operatively and then one week, two weeks, four weeks, three months, six months, and one year post-operatively. Patient clinical outcomes will be captured using web-based progress reports. Patients will complete the Quality of Life (QoL-12), Neck Disability Index (NDI), and Visual Analog Scale (VAS) questionnaires electronically pre-operatively and at one year post-operatively. This outcome data will help us analyze the swallowing function or symptoms with the overall clinical course of the patients enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Elective anterior approach to subaxial cervical spine (C3 - T1);
* ages 18-80

Exclusion Criteria:

* Traumatic or tumor etiologies
* undergoing anterior-posterior operations
* neoplastic, or infectious conditions requiring surgery
* a history of previous anterior cervical spine surgery
* any patient requiring a halo vest
* patients on chronic steroids
* patients remaining intubated post-operatively (please see more under risks below)
* less than 18 years of age
* pregnant women
* no phone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-07; Primary Completion 2016-05-15 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanford E Emery, MD, MBA, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Group data will be available via publication. Participants are told their randomization assignment at one year, or up to two year, follow up post surgery, dependent on their return to clinic.
Supporting Information: Study Protocol
Time Frame: Within one year of study completion
Access Criteria: Through a published manuscript and to participants via phone call or clinic visit when the participants return for regularly scheduled follow up visits.

REFERENCES:
- [Background] Riley LH 3rd, Vaccaro AR, Dettori JR, Hashimoto R. Postoperative dysphagia in anterior cervical spine surgery. Spine (Phila Pa 1976). 2010 Apr 20;35(9 Suppl):S76-85. doi: 10.1097/BRS.0b013e3181d81a96. PMID 20407354
- [Background] Fountas KN. Re: Papavero L, Heese O, Klotz-Regener V, et al. The impact of esophagus retraction on early dysphagia after anterior cervical surgery. Spine 2007;32:1089-93. Spine (Phila Pa 1976). 2007 Dec 15;32(26):3090. doi: 10.1097/BRS.0b013e31815cd40f. No abstract available. PMID 18091507
- [Background] Mendoza-Lattes S, Clifford K, Bartelt R, Stewart J, Clark CR, Boezaart AP. Dysphagia following anterior cervical arthrodesis is associated with continuous, strong retraction of the esophagus. J Bone Joint Surg Am. 2008 Feb;90(2):256-63. doi: 10.2106/JBJS.G.00258. PMID 18245583
- [Background] Cavusoglu H, Tuncer C, Tanik C, Mutlu Z, Zengin E, Karabagli M, Aydin Y. The impact of automatic retractors on the esophagus during anterior cervical surgery: an experimental in vivo study in a sheep model. J Neurosurg Spine. 2009 Nov;11(5):547-54. doi: 10.3171/2009.6.SPINE09216. PMID 19929356
- [Background] Lee MJ, Bazaz R, Furey CG, Yoo J. Risk factors for dysphagia after anterior cervical spine surgery: a two-year prospective cohort study. Spine J. 2007 Mar-Apr;7(2):141-7. doi: 10.1016/j.spinee.2006.02.024. Epub 2007 Jan 22. PMID 17321961
- [Background] Rihn JA, Kane J, Albert TJ, Vaccaro AR, Hilibrand AS. What is the incidence and severity of dysphagia after anterior cervical surgery? Clin Orthop Relat Res. 2011 Mar;469(3):658-65. doi: 10.1007/s11999-010-1731-8. PMID 21140251
- [Background] Siska PA, Ponnappan RK, Hohl JB, Lee JY, Kang JD, Donaldson WF 3rd. Dysphagia after anterior cervical spine surgery: a prospective study using the swallowing-quality of life questionnaire and analysis of patient comorbidities. Spine (Phila Pa 1976). 2011 Aug 1;36(17):1387-91. doi: 10.1097/BRS.0b013e31822340f2. PMID 21785303
- [Background] Kang SH, Kim DK, Seo KM, Kim KT, Kim YB. Multi-level spinal fusion and postoperative prevertebral thickness increase the risk of dysphagia after anterior cervical spine surgery. J Clin Neurosci. 2011 Oct;18(10):1369-73. doi: 10.1016/j.jocn.2011.02.033. Epub 2011 Jul 27. PMID 21798743
- [Background] Bazaz R, Lee MJ, Yoo JU. Incidence of dysphagia after anterior cervical spine surgery: a prospective study. Spine (Phila Pa 1976). 2002 Nov 15;27(22):2453-8. doi: 10.1097/00007632-200211150-00007. PMID 12435974
- [Background] Riley LH 3rd, Skolasky RL, Albert TJ, Vaccaro AR, Heller JG. Dysphagia after anterior cervical decompression and fusion: prevalence and risk factors from a longitudinal cohort study. Spine (Phila Pa 1976). 2005 Nov 15;30(22):2564-9. doi: 10.1097/01.brs.0000186317.86379.02. PMID 16284596
- [Background] Pedram M, Castagnera L, Carat X, Macouillard G, Vital JM. Pharyngolaryngeal lesions in patients undergoing cervical spine surgery through the anterior approach: contribution of methylprednisolone. Eur Spine J. 2003 Feb;12(1):84-90. doi: 10.1007/s00586-002-0495-6. Epub 2002 Dec 4. PMID 12592551
- [Background] Emery SE, Akhavan S, Miller P, Furey CG, Yoo JU, Rowbottom JR, Bohlman HH. Steroids and risk factors for airway compromise in multilevel cervical corpectomy patients: a prospective, randomized, double-blind study. Spine (Phila Pa 1976). 2009 Feb 1;34(3):229-32. doi: 10.1097/BRS.0b013e318193a287. PMID 19148042
- [Background] Lee SH, Kim KT, Suk KS, Park KJ, Oh KI. Effect of retropharyngeal steroid on prevertebral soft tissue swelling following anterior cervical discectomy and fusion: a prospective, randomized study. Spine (Phila Pa 1976). 2011 Dec 15;36(26):2286-92. doi: 10.1097/BRS.0b013e318237e5d0. PMID 22020609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants undergoing elective anterior cervical spine surgery will be seen by spine surgeons at the WVU Spine Center. Participants will be told about the study and given the opportunity to consent. Consented participants will be randomized to either the steroid administration group or the saline administration group.
Groups:
- Treatment 1; Dexamethasone: Swallowing difficulty at various time points as measured by the DSQ and Bazaz for subjects randomized to Treatment 1; Dexamethasone
- Treatment 0; Saline Placebo: Swallowing difficulty at various time points as measured by the DSQ and Bazaz for subjects randomized to Treatment 0; Saline placebo
Period: Overall Study
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Saline Placebo
Started | 36 | 38
Double Blind (0-52 Weeks) | 36 | 38
Last Participant Completed 1 yr | 33 | 31
Completed | 33 | 31
Not Completed | 3 | 7
Not completed — given steroids | 1 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — recruited during continuing renewal proc | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — surgery started late | 0 | 1
Not completed — re-operation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Ten participant's data was not analyzed for various reasons.
Groups:
- Treatment 1; Dexamethasone: Patients undergoing elective anterior cervical spine surgery will be seen by spine surgeons. After consent the Bazaz and Dysphagia Short Questionnaire will be administered at baseline prior to surgery, Day 1, Day 2, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  Patients will be randomized to either the steroid administration group or the saline administration group. Patients randomized to the experimental (steroid) group will receive 0.3 mg/kg of intravenous dexamethasone within one hour of the incision, then 0.15 mg/kg every eight hours for two doses. This dosage is approximately 20 mg, 10 mg, and 10 mg of dexamethasone. Patients in the control(saline) group will receive a similar volume of saline on the same schedule for three doses.
  Treatment 1; Dexamethasone: Dexamethasone IV given within the first hour of surgery; second dose given 8 hours after first dose; third dose given 8 hours after second dose.
- Treatment 0; Saline Placebo: Patients undergoing elective anterior cervical spine surgery will be seen by spine surgeons. After consent the Bazaz and Dysphagia Short Questionnaire will be administered at baseline prior to surgery, Day 1, Day 2, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  Patients will be randomized to either the steroid administration group or the saline administration group. Patients randomized to the experimental (steroid) group will receive 0.3 mg/kg of intravenous dexamethasone within one hour of the incision, then 0.15 mg/kg every eight hours for two doses. This dosage is approximately 20 mg, 10 mg, and 10 mg of dexamethasone. Patients in the control(saline) group will receive a similar volume of saline on the same schedule for three doses.
  Treatment 0; Saline placebo: Saline (placebo) IV given within the first hour of surgery; second dose given 8 hours after first dose; third dose given 8 hours after second dose.
- Total: Total of all reporting groups
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Saline Placebo | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Categorical [Count of Participants; unit: Participants] — Population: Ten total subjects were removed from the study for various reasons.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 30 | 31 | 61
    >=65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 13 | 15 | 28
Region of Enrollment [Number; unit: participants] — The Dysphagia Short Questionnaire: An Instrument for Evaluation of Dysphagia (DSQ) and Bazaz Dysphagia Scale (Bazaz) were administered in person at baseline and Day 1, via phone call Day 2, Week 1,2; 1,3, 6 months, and 1 year.
  participants
    United States | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Swallowing Difficulty
Description: Two measurement surveys were used: The Dysphagia Short Questionnaire: An Instrument for Evaluation of Dysphagia (DSQ) and Bazaz Dysphagia Scale (Bazaz). The DSQ and Bazaz determine levels of dysphagia over time after anterior cervical spine surgery. A DSQ score of zero indicates no symptoms. Any number above zero indicates difficulty swallowing. The Bazaz score of Zero indicates no symptoms. Any number above zero indicates difficulty swallowing. Numbers of subjects reporting any difficulty swallowing (had to have a score of at least 1) at various time points are listed below associated with the randomization assignment and survey used.
Time Frame: 1 day; 2 days; 1 week; 2 weeks; 1 month; 3 months; 6 months;12 months
Population: Treatment 1; Dexamethasone or Treatment 0; Saline placebo. Treatment 1 received 0.3 mg/kg of intravenous dexamethasone within one hour of the incision, then 0.15 mg/kg every eight hours for two doses. Dosage was approximately 20 mg, 10 mg, and 10 mg of dexamethasone. Treatment 0 received similar volume of saline on same schedule for three doses.
Measure: Count of Participants; unit: Participants
Groups:
- Dexamethasone DSQ: Treatment 1; Dexamethasone. Patients undergoing elective anterior cervical spine surgery were seen by spine surgeons. After consent the Bazaz and Dysphagia Short Questionnaire were administered at baseline prior to surgery, Day 1, Day 2, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  Patients were randomized to either the steroid administration group or the saline administration group. Patients randomized to the experimental (steroid) group received 0.3 mg/kg of intravenous dexamethasone within one hour of the incision, then 0.15 mg/kg every eight hours for two doses. This dosage is approximately 20 mg, 10 mg, and 10 mg of dexamethasone.
  Treatment 1; Dexamethasone: Dexamethasone IV given within the first hour of surgery; second dose given 8 hours after first dose; third dose given 8 hours after second dose.
- Saline Placebo DSQ: Treatment 0; Saline Placebo. Patients undergoing elective anterior cervical spine surgery wereseen by spine surgeons. After consent the Bazaz and Dysphagia Short Questionnaire were administered at baseline prior to surgery, Day 1, Day 2, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  Patients were randomized to either the steroid administration group or the saline administration group. Patients randomized to the control (saline) group received 0.3 mg/kg of intravenous saline within one hour of the incision, then 0.15 mg/kg every eight hours for two doses. This dosage is approximately 20 mg, 10 mg, and 10 mg of saline.
  Treatment 0; Control (Saline) IV given within the first hour of surgery; second dose given 8 hours after first dose; third dose given 8 hours after second dose.
- Dexamethasone Bazaz: Treatment 1; Dexamethasone. Treatment 1; Dexamethasone. Patients undergoing elective anterior cervical spine surgery were seen by spine surgeons. After consent the Bazaz and Dysphagia Short Questionnaire were administered at baseline prior to surgery, Day 1, Day 2, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  Patients were randomized to either the steroid administration group or the saline administration group. Patients randomized to the experimental (steroid) group received 0.3 mg/kg of intravenous dexamethasone within one hour of the incision, then 0.15 mg/kg every eight hours for two doses. This dosage is approximately 20 mg, 10 mg, and 10 mg of dexamethasone.
  Treatment 1; Dexamethasone: Dexamethasone IV given within the first hour of surgery; second dose given 8 hours after first dose; third dose given 8 hours after second dose.
- Saline Placebo Bazaz: Treatment 0; Saline Placebo. Treatment 0; Saline Placebo. Patients undergoing elective anterior cervical spine surgery wereseen by spine surgeons. After consent the Bazaz and Dysphagia Short Questionnaire were administered at baseline prior to surgery, Day 1, Day 2, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  Patients were randomized to either the steroid administration group or the saline administration group. Patients randomized to the control (saline) group received 0.3 mg/kg of intravenous saline within one hour of the incision, then 0.15 mg/kg every eight hours for two doses. This dosage is approximately 20 mg, 10 mg, and 10 mg of saline.
  Treatment 0; Control (Saline) IV given within the first hour of surgery; second dose given 8 hours after first dose; third dose given 8 hours after second dose.
Arm/Group | Dexamethasone DSQ | Saline Placebo DSQ | Dexamethasone Bazaz | Saline Placebo Bazaz
Number analyzed (Participants) | 33 | 31 | 33 | 31
Participants
  Difficulty swallowing Baseline | 16 | 14 | 5 | 7
  Difficulty swallowing day 1 | 24 | 28 | 19 | 21
  Difficulty swallowing day 2 | 22 | 28 | 15 | 23
  Difficulty swallowing Week 1 | 29 | 28 | 14 | 21
  Difficulty swallowing Week 2 | 23 | 27 | 14 | 19
  Difficulty swallowing Month 1 | 19 | 24 | 13 | 17
  Difficulty swallowing Month 3 | 9 | 17 | 3 | 11
  Difficulty swallowing Month 6 | 6 | 11 | 2 | 10
  Difficulty swallowing Month 12 | 11 | 13 | 7 | 8
Statistical Analysis 1: Comparison: Dexamethasone DSQ vs Saline Placebo DSQ; Comparing DSQ between Dexamethasone and Saline at Day 1 post-op; Test type: Superiority; p = 0.036, t-test, 2 sided; Mean Difference (Final Values) = -1.5392, 95% CI 2-sided [-2.9761 to -.1022], Standard Error of Mean .7176
Statistical Analysis 2: Comparison: Dexamethasone Bazaz vs Saline Placebo Bazaz; Comparing Bazaz between Dexamethasone and Saline at 6 months post-op; Test type: Superiority; p < .05, t-test, 2 sided; Mean Difference (Final Values) = -.6040, 95% CI 2-sided [-1.1151 to -.0930], Standard Error of Mean .2543

2. Secondary Outcome: Change in Quality of Life
Description: Change in Quality of life measured by the Neck Disability Index (NDI) from baseline and 1 year for Treatment 1; Dexamethasone and Treatment 0; Saline placebo. The NDI measures self-rated disability due to neck pain. Each of the 10 items is scored from 0 - 5. The maximum score is 50. The higher the score the more disability. The scale is 0 - 4 = no disability; 5 - 14 = mild;15 - 24 = moderate; 25 - 34 = severe; above 34 = complete disability.
Time Frame: Baseline and 1 year (or last visit as appropriate). Not all subjects followed up at 1 year.
Population: Neck Disability Index change from baseline to 1 year or last visit as appropriate. Not all subjects followed up at 1 year.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Change in Quality of Life Dexamethasone: Change in quality of life from baseline to 1 year (or last visit as appropriate). Not all subjects came for 1 year follow up.
- Change in Quality of Life Saline Placebo: Change in quality of life from baseline to 1 year (or last visit as appropriate.) Not all subjects came for 1 year follow up.
Arm/Group | Change in Quality of Life Dexamethasone | Change in Quality of Life Saline Placebo
Number analyzed (Participants) | 33 | 31
units on a scale | -6.1208 (3.1273) | -7.9082 (3.1273)
Statistical Analysis 1: Comparison: Change in Quality of Life Dexamethasone vs Change in Quality of Life Saline Placebo; Comparing the changes in VNDI between Dexamethasone and Saline from baseline to last visit; Test type: Superiority; p < .05, t-test, 2 sided; Mean Difference (Final Values) = 1.7874, 95% CI 2-sided [-4.5153 to 8.0902], Standard Error of Mean 3.1273

3. Secondary Outcome: Fusion Rate Steroid vs Placebo
Description: Participants were considered fused if radiographs demonstrated less than 1 millimeter of interspinous motion between flexion and extension,7 or if CT/MRI demonstrated clear evidence of bone bridging from endplate to endplate.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Dexamethasone Fusion; Saline Fusion: Fused if radiographs demonstrated less than 1 millimeter of interspinous motion between flexion and extension,7 or if CT/MRI demonstrated clear evidence of bone bridging from endplate to endplate.
Arm/Group | Dexamethasone Fusion | Saline Fusion
Number analyzed (Participants) | 33 | 31
Participants
  unknown | 13 | 19
  fused | 20 | 11
  not fused | 0 | 1
Statistical Analysis 1: Comparison: Dexamethasone Fusion vs Saline Fusion; Test type: Superiority; p = .375, Fisher Exact — Fisher's Exact Test

ADVERSE EVENTS:
Time Frame: up to 1 year
Description: Other not including serious adverse events
Groups:
- Treatment 1; Dexamethasone; Treatment 0; Saline Placebo: Swallowing difficulty. Two measurement surveys were used: The Dysphagia Short Questionnaire: An Instrument for Evaluation of Dysphagia (DSQ) and Bazaz Dysphagia Scale (Bazaz). The DSQ and Bazaz determine levels of dysphagia over time after anterior cervical spine surgery. A DSQ score is calculated by summing up the points given for each item to a maximum of 18 points, where lower scores represent milder symptoms (zero indicates no symptoms) and vice versa. For the Bazaz score, symptoms are measured as 'none', 'mild', 'moderate', or 'severe'. Zero indicates none or no symptoms, 1 indicates mild, 2 indicates moderate, 3 indicates severe. Numbers of subjects reporting any difficulty swallowing (had to have a score of at least 1) at various time points are reported.
Arm/Group | Treatment 1; Dexamethasone | Treatment 0; Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 0/33 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1; Dexamethasone (N=33) | Treatment 0; Saline Placebo (N=31)
intraoperative musculoskeletal injury (Surgical and medical procedures) | 0 (0) | 0 (0)
intraoperative neurological injury (Surgical and medical procedures) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2014-05-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT02416934/Prot_000.pdf